CLINICAL TRIAL: NCT04135898
Title: A Randomized, Double-blind, Phase I Study Comparing the Pharmacokinetic and Safety of SIBP-04 and Bevacizumab in Healthy Male Subjects
Brief Title: A Study Comparing SIBP-04 and Bevacizumab in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIBP-04-01
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Healthy Male
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIBP-04 (Experimental)
  Interventions: Drug: SIBP-04
- Bevacizumab (Active Comparator)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: SIBP-04 — 3mg/kg, infusion in 90 minutes
  Arms: SIBP-04
Drug: Bevacizumab — 3mg/kg, infusion in 90 minutes
  Arms: Bevacizumab

SUMMARY:
This is a randomised, double-blind, positive drug parallel controlled clinical trial in China. In the trial, it is planned to enroll 88 subjects, randomized to two treatment groups in a ratio of 1:1 to receive the test drug and the positive control.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able and willing to give written informed consent.
2. 18-45 years old, male.
3. Body mass index (BMI): 18-26 kg/m2 (including 18 kg/m2 and 26 kg/m2), and weighing between 50-80 kg (including 50 kg and 80 kg).
4. Subjects determined healthy by Vital signs, physical examination, laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, fecal occult blood, etc.), 12-lead electrocardiogram, chest X-ray, abdominal ultrasound, urinary ultrasound, without any clinically significant abnormality judged by the investigator.
5. Subjects who are willing to comply with the contraception restrictions from signing of the informed consent form until 6 months after the infusion of the test drug.
6. Subjects who can participate in the visit on time and complete the visit.

Exclusion Criteria:

1. Subjects with the following diseases, including but not limited to: nervous system, cardiovascular system, blood and lymphatic system, immune system, digestive system, respiratory system, metabolism and bone diseases.
2. History of digestive tract perforation or digestive tract disease.
3. Subjects who are allergic to Avastin® and its ingredients.
4. History of autoimmune diseases or allergic diseases.
5. History of clinically significant proteinuria (urine routine examination, urinary protein 2+and above) or proteinuria judged by the investigator.
6. Any inherited predisposition to bleeding or to thrombosis or history of non traumatic hemorrhage (i.e., requiring medical intervention), thromboembolic event or any condition which may increase bleeding risk including clotting disorders, thrombocytopenia (platelet count < 125000/µL) or an international normalized ratio (INR) higher than 1.5.
7. Subjects who did strenuous exercise 96 hours before the test, or participate in intense physical activity within 30 days after the scheduled dose, including physical contact or impact sports;
8. Subject with a family history of cancer or a malignant tumor within the past 5 years.
9. Abnormal ECG with clinical significance judged by the Investigator.
10. Subjects with relevant family history of hypertension or abnormal blood pressure at screening or admission to the study center (Day 1): (Systolic blood pressure ≤ 90mmHg or ≥ 140mmHg, or / and diastolic blood pressure ≤ 60mmHg or ≥ 90mmHg), heart rate ≤ 50bpm or ≥ 100bpm.
11. Subjects who have acute or chronic infectious diseases and have clinical significance during the screening and admission studies, or hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), hepatitis B surface antigen (HBsAg), syphilis test positive during the screening.
12. History of prior exposure to bevacizumab or any anti VEGF monoclonal antibodies or proteins.
13. Live virus vaccination within 3 months prior to study drug administration， or prior exposure to any other investigational monoclonal antibody within 9 months.
14. Intake of prescribed or over the counter drugs within 5 half-life of the drug or 2 weeks prior to the use of the test drug, or intake of herbal drugs or dietary supplements within 28 days prior to randomization.
15. Use of any investigational drug in any clinical study within the 3 months prior to Sign informed consent.
16. Blood loss or blood donation (including blood components donation) ≥ 400 mL or blood transfusion within 3 months before study drug administration.
17. Unhealed wound ulcers or fractures, or major surgery within 2 months prior to randomization or expected major surgery during the study period or 2 months after the end of the study.
18. Plan to receive oral or dental surgery during the study period.
19. History of alcohol abuse or a positive alcohol breath test before study drug administration.
20. History of drug abuse, or have positive drug screening results.
21. Subjects who have more than 5 cigarettes per day within 3 months before enrollment.
22. Others that are not in compliance with the enrollment judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
AUC0-t | From 0 to day 71
  Area under the concentration time curve of the analyte in serum over the time interval from 0 to the last measurable concentration at time "t"

SECONDARY OUTCOMES:
Cmax | From 0 to day 71
  Maximum measured concentration of the analyte in serum
AUCinf | From 0 to day 71
  Area under the concentration time curve of the analyte in serum over the time interval from 0 to extrapolated to infinite time
Tmax | From 0 to day 71
  Time from dosing to maximum measured concentration
t1/2 | From 0 to day 71
  Terminal half life of the analyte in serum
λz | From 0 to day 71
  Terminal elimination rate constant
CL | From 0 to day 71
  Total clearance of the analyte in serum following IV infusion
Vd | From 0 to day 71
  Volume of distribution during the terminal phase λz following an intravascular dose
Immunogenicity | From 0 to day 71
  Incidence of anti drug antibodies (ADAs) and neutralizing anti drug antibodies（NAb）

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai Institute Of Biological Products Co., Ltd, Study Director — SINOPHARM; The First Affiliated Hospital, Principal Investigator — Bengbu Medical College
Locations (1):
- the First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China